CLINICAL TRIAL: NCT05746533
Title: A Comparison of Total Hip Arthroplasty and Hip Preservation Outcomes
Brief Title: An Evaluation of Hip Preservation Outcomes
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2000032269
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hip Arthroscopy; Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants Undergoing Hip Preservation/Surgical Interventions: Data will be prospectively collected on participants undergoing hip preservation at Yale-New Haven Hospital.
  Interventions: Procedure: Hip Arthroscopy

INTERVENTIONS:
Procedure: Hip Arthroscopy — Hip Preservation surgeries

SUMMARY:
The purpose of this study is to assess outcomes of hip preservation surgeries including open and arthroscopic treatment of femoroacetabular impingement (FAI).

DETAILED DESCRIPTION:
The purpose of this study is to assess outcomes of hip preservation surgeries including open and arthroscopic treatment of femoroacetabular impingement (FAI). Data will be prospectively and retrospectively collected on about 10,000 patients undergoing hip preservation at Yale-New Haven Hospital. Patients who are candidates for surgical intervention of the hip are potential participants.

The primary objective of this study is to determine whether hip arthroscopy reduces or improves post-operative outcome measures compared to pre-operative measures (including patient reported outcomes [PROs], revision surgery, conversion to total hip arthroplasty, and return to sport) in patients with FAI and labral tears.

The secondary objective of this study is to be able to better gauge (by assessments of patient satisfaction and psychometric thresholds of success) the progress made by recent advancements in arthroscopic hip preservation procedures with longitudinal follow-up.

The focus of this clinical trial will be the data collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for surgical intervention of the hip
* Participant and/or guardian has given informed consent and assent as applicable.

Exclusion Criteria:

* Documented history of pre-existing hip conditions (SCFE, LCPD, acetabular fractures)
* Has language or cognitive barriers preventing understanding of study and consent and assent documents
* Prior revision surgeries
* Patients from the trauma/emergency department
* Individuals with Unusable x-rays

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients age 12 years and older who are candidates for surgical intervention of the hip.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2053-06 (Estimated); Study Completion 2053-06 (Estimated)

PRIMARY OUTCOMES:
Change in Hip Outcome Score (iHOT-12) | Baseline, 3 months post-operatively, 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
  iHOT-12 is a 12-item questionnaire scored using a visual analog scale from 0 to 100, with a score of 100 being the best function and least amount of symptoms, and the overall mean equates to the final iHOT score.
Change in Hip Outcome Score (HOS) | Baseline, 3 months post-operatively, 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
  The HOS is a self-administered questionnaire with a scoring system composed of 2 sub-scales. The 19 item Activities of Daily Living (ADL) sub-scale and a 9 item Sports sub-scale. Both have a range of scores from 0 to 4, with 0 being 'unable to do' and 4, 'no difficulty'. N/A is also an option. The total score for each is multiplied by 4 with the highest potential ADL score bing no greater than 68 and the sports scale with the highest potential score being 36. An overall higher score from both sub-scales indicates a greater level of function.
Change in PROMIS questionnaire Score | Baseline, 3 months post-operatively, 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
  PROMIS Physical function is a standardized computer adapted test which is able to quickly and effectively score patients on a scale of 0 (not able to function) to 100 (fully functional) based on their physical function. 100 would be a perfect score and 0 would be the worst possible score. Higher scores indicate better physical function.
Change in Sports Survey Score | Baseline, 3 months post-operatively, 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
  The Chicago sports score asks athletes questions pertaining to their ability to return to sport. If they are able to return to sport it asks questions about their ability level since returning. Similarly, if they are not able to return to sport it asks questions regarding what has held them back. It is on a 100 point scale with 100 being the best possible outcome and 0 the lowest possible score. Higher scores indicate better ability to return to sports.
Change in Pain Score using a visual analog scale (VAS) | Baseline, 3 months post-operatively, 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
  Participants will be asked to estimate their pain on a VAS from 0 to 10, where 0 is considered to be no pain at all and 10 is considered to be the worst possible pain.
Change in PROMIS Pain Interference | Baseline, 3 months post-operatively, 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
  Participants will receive the PROMIS pain interference, physical function, and global health modules to assess quality of life, a commonly used general health quality of life assessment tool. PROMIS pain interference is a standardized computer adapted test which is able to quickly and effectively score patients on a scale of 0-100 based on how pain affects their day to day life. 100 would be a perfect score and 0 would be the worst possible score. Higher scores indicate less pain interference on quality of life.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 | Baseline, 3 months post-operatively, 6 months post-operatively, 1 year post-operatively, 2 years post-operatively, 5 years post-operatively, and 10 years post-operatively
  The PROMIS Global-10 is a 10-item patient-reported questionnaire that measures changes in general health in which the response options are presented as 5-point scale, 5 (without any difficulty) to 1 (Unable to do). Higher scores indicate a healthier patient.

SECONDARY OUTCOMES:
Change in Patients Satisfaction Post Surgery | 3 months, 6 months, 1 year, 2 year, 5 year and 10 year
  Participants will be asked to rate their level of satisfaction after surgery with 10 being extremely satisfied and 0 being not satisfied at all.
Psychometric thresholds of success will be assessed using anchor questions | up to 10 years
  Participants will be asked anchor questions which will be used to determine psychometric thresholds of success the psychometric threshold substantial clinical benefit (SCB). They will be asked whether they feel that their current symptoms are acceptable or not to them. This helps to establish the patient acceptable symptomatic state (PASS). They will also be asked whether they feel that their hip is better worse or no different compared to before surgery. This will establish the psychometric threshold SCB.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Jimenez, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant outcomes and demographic data will be shared with other researchers for the purpose of collaboration.
Supporting Information: CSR
Time Frame: Beginning 12 months and ending 36 months following primary publication.
Access Criteria: Proposals should be directed to andrew.jimenez@yale.edu. To gain access, data requestors may need to sign a data use access/use agreement and have approval from an institutional review board/ethics board for the proposed use of such data.